CLINICAL TRIAL: NCT03455660
Title: A Retrospective Comparison of Neonatal Acid-base Status After Cesarean Delivery (CD) at NYPresbyterian/Columbia University Medical Center (CUMC) Before January, 2015 and After January, 2016
Brief Title: A Retrospective Comparison of Neonatal Acid-base Status After CD Before January, 2015 and After January, 2016
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Allison Lee, Assistant Professor of Anesthesiology, Columbia University
Other Study IDs: AAAR7164
Record Dates: First submitted 2018-01-04; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Cesarean Delivery
Keywords: Cesarean; C-Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-January 2015: Patients who underwent cesarean delivery between February 2013 and December 2014.
  Interventions: Other: no intervention
- Post-January 2016: Patients who underwent cesarean delivery between February 2016 and December 2017.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The objective is to retrospectively gather peri-operative data on neonatal outcomes, primarily neonatal acid-base status, based on umbilical cord gas analysis, for the 23 months preceding and 23 months following the conduct of the "tilt versus supine study". The investigators hypothesize that there will be no difference in mean neonatal umbilical artery base excess in neonates delivered by cesarean section during the period before and after conduct of the study, for elective, urgent and emergent deliveries.

DETAILED DESCRIPTION:
For decades, obstetric anesthesia dogma for term women undergoing cesarean delivery (CD) includes maintenance of left lateral tilt for uterine displacement until delivery, based on the premise that the supine position will result in aortocaval compression (ACC), maternal hypotension and fetal compromise. More recent evidence suggests that even in 15 degrees of left tilt, there is minimal relief of aortocaval compression. Furthermore, there is evidence that most practitioners never achieve 15 degrees of tilt anyway.

Between January 2015 and January 2016, the investigators conducted a randomized clinical trial at NewYork Presbyterian/The Allen Hospital in which healthy women undergoing elective CD were randomized (non-blinded) to supine horizontal (SUPINE, N=50) or 15° left tilt of the surgical table (TILT, N= 50) following spinal anesthesia (hyperbaric bupivacaine 12 mg, fentanyl 15 μg, preservative-free morphine 150 μg). Lactated Ringer's 10ml/kg and a phenylephrine (PE) infusion titrated to 100% baseline systolic blood pressure (SBP) were initiated with intrathecal injection. The primary outcome was umbilical artery base excess (UA-BE). There were no differences in UA-BE or pH between groups. The mean UA-BE (± SD) was -0.5 mmol/L (± 1.6) in the SUPINE group (n=50) versus -0.6 mmol/L (± 1.5) in the TILT group (n=47) (p= 0.64). The conclusion was that maternal supine position during elective CD with spinal anesthesia in healthy term women does not impair neonatal acid-base status compared to 15° left tilt, when maternal SBP is maintained with a coload and PE infusion. The investigators understood that the findings may not be generalized to emergency situations or non-reassuring fetal status.

Since the end of the study, discussion of the findings with colleagues at Departmental grand rounds and national conferences, and a publication in the journal Anesthesiology, practitioners have reported feeling more comfortable with maternal supine position during cesarean delivery, as long as maternal SBP is kept at or near to baseline with crystalloid infusion and a PE infusion. It is routine practice at CUMC to use a prophylactic PE infusion for maintenance of maternal SBP close to or at baseline. It is also routine at CUMC to send samples of umbilical arterial and venous blood for analysis. Much of the dosing for neuraxial anesthesia (spinal, combined spinal epidural anesthesia and epidural doses) are standardized at CUMC. The investigators believe that since there has been a noticeable practice shift with practitioners anecdotally reporting that they have discontinued the routine use of left maternal tilt intraoperatively, the investigators will be able to collect useful data on cases which had not been studied - these include cases with preeclampsia, morbid obesity and emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Women who delivered between February 2013 and December 2014, and between February 2016 and December 2017

Exclusion Criteria:

* none

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Retrospective cohorts of women who delivered between February 2013 and December 2014, and between February 2016 and December 2017
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Umbilical artery base excess | 10 minutes
  Base excess calculation of umbilical artery blood

SECONDARY OUTCOMES:
Umbilical artery pH | 10 minutes
  pH measurement of umbilical artery blood

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lee, MD, Principal Investigator — Columbia University
Locations (1):
- NewYork Presbyterian/The Allen Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Will not share patient identifiable data with other researchers.

REFERENCES:
- [Background] Lee AJ, Landau R. Aortocaval Compression Syndrome: Time to Revisit Certain Dogmas. Anesth Analg. 2017 Dec;125(6):1975-1985. doi: 10.1213/ANE.0000000000002313. PMID 28759487
- [Background] Higuchi H, Takagi S, Zhang K, Furui I, Ozaki M. Effect of lateral tilt angle on the volume of the abdominal aorta and inferior vena cava in pregnant and nonpregnant women determined by magnetic resonance imaging. Anesthesiology. 2015 Feb;122(2):286-93. doi: 10.1097/ALN.0000000000000553. PMID 25603203
- [Background] Jones SJ, Kinsella SM, Donald FA. Comparison of measured and estimated angles of table tilt at Caesarean section. Br J Anaesth. 2003 Jan;90(1):86-7. PMID 12488385
- [Background] Aust H, Koehler S, Kuehnert M, Wiesmann T. Guideline-recommended 15 degrees left lateral table tilt during cesarean section in regional anesthesia-practical aspects: An observational study. J Clin Anesth. 2016 Aug;32:47-53. doi: 10.1016/j.jclinane.2015.12.041. Epub 2016 Mar 22. PMID 27290944
- [Background] Lee AJ, Landau R, Mattingly JL, Meenan MM, Corradini B, Wang S, Goodman SR, Smiley RM. Left Lateral Table Tilt for Elective Cesarean Delivery under Spinal Anesthesia Has No Effect on Neonatal Acid-Base Status: A Randomized Controlled Trial. Anesthesiology. 2017 Aug;127(2):241-249. doi: 10.1097/ALN.0000000000001737. PMID 28598894